CLINICAL TRIAL: NCT02266147
Title: A Phase 1/2, Non-randomized, Open-label, Multicenter, Dose Escalation and Expansion Study of Intratumoral Injections of SD-101 in Combination With Localized Low-dose Radiation in Patients With Untreated Low-grade B-cell Lymphoma
Brief Title: Study of SD-101 in Combination With Localized Low-dose Radiation in Patients With Untreated Low-grade B-cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor terminated the trial early because there was sufficient data to make a decision about SD-101 in the lymphoma development program.
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DV3-LYM-01
Record Dates: First submitted 2014-10-13; First posted 2014-10-16 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: B-cell Lymphoma
Keywords: Low Grade B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SD-101 in combination with low-dose radiation (Experimental): PART 1
  * Radiation: 2 fractions of 2 Gy over 2 days at Days -1 and 1
  * COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29
  * COHORT 2: 2 mg/mL at Days 1, 8, 15, 22, and 29
  * COHORT 3: 4 mg/mL at Days 1, 8, 15, 22, and 29
  * COHORT 4: 8 mg/mL at Days 1, 8, 15, 22, and 29
  PART 2
  Cycle 1: Required
  * Radiation: 2 fractions of 2 Gy over 2 days at Days -1 and 1
  * COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29
  * COHORT 2: 8 mg/mL at Days 1, 8, 15, 22, and 29
  Cycle 2: Optional
  * Radiation: 2 fractions of 2 Gy over 2 days at Days 180 and 181
  * COHORT 1: 1 mg/mL at Days 181, 188, 195, 202, and 209
  * COHORT 2: 8 mg/mL at Days 181, 188, 195, 202, and 209
  Interventions: Drug: SD-101; Radiation: Radiation therapy

INTERVENTIONS:
Drug: SD-101
Radiation: Radiation therapy

SUMMARY:
To assess the safety and tolerability of escalating doses of SD-101 in combination with localized low-dose radiation therapy in adult subjects with untreated low-grade B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed, untreated, low-grade B-cell lymphoma, including follicular (Grade 1, 2, or 3A) [Harris, Swerdlow et al. 2008] or marginal, or CLL/SLL with lymph node involvement.
* At least 2 sites of measurable disease per Cheson criteria (must measure at least 1.5 cm in any diameter or 1.0 cm in the shortest diameter if one of the diameters is not ≥ 1.5 cm), one of which must be palpable and easily accessible in a low-risk site (eg, inguinal, axillary, cervical, subcutaneous) for intratumoral injection (denoted as "Lesion A" in Treatment Cycle 1) and at least one additional untreated lesion that is located outside the radiation field of the treated lesion (Lesion A) and is accessible for an FNA aspirate.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Aged 18 years and older
* Absolute neutrophil count (ANC) ≥ 1500/mm3
* Platelet count > 100,000/µL
* Serum creatinine (Cr) ≤ 1.5 x upper limit of normal (ULN).
* Serum total bilirubin ≤ 1.5 x the ULN.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* International normalized ratio or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy and the PT or partial thromboplastin time (PTT) must be within the therapeutic range of the intended use of anticoagulants.
* Activated PTT (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy, and the PT or PTT is within therapeutic range of intended use of anticoagulants.
* Female subjects must have a negative urine or serum pregnancy test within 72 hours prior to taking study medication if of childbearing potential as defined in this protocol. Women of childbearing potential (WOCBP) must be willing to use 2 medically acceptable method of contraceptive from Day 1 through 120 days after the last dose of trial treatment. The 2 medically acceptable birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), cooper intrauterine device, sponge, or spermicide as per local regulations or guidelines. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
* Ability to understand and sign informed consent form (ICF) and comply with treatment protocol

Exclusion Criteria:

* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy (including immune modulators or systemic corticosteroids) within 7 days prior to study enrollment.
* Positive for hepatitis B (HBsAg reactive), HCV ribonucleic acid (RNA) qualitative, or human immunodeficiency virus (HIV)( HIV 1/2 antibodies)
* Diagnosis of mantle or diffuse large-cell lymphoma, Grade 3B follicular lymphoma [Harris, Swerdlow et al. 2008] or gastric mucosa-associated lymphoid tissue (MALT) lymphoma
* Clinically significant pleural effusion
* Active infection including cytomegalovirus
* Pregnant or breast feeding within the projected duration of trial participation through 4 months after the last dose of study treatment.
* Autoimmune disease including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjӧgren's syndrome, autoimmune thrombocytopenia, history of uveitis, or other if clinically significant
* Lymphoma involvement of the central nervous system
* Received any prior therapy for lymphoma
* Use of any investigational agent within the last 28 days
* Serious, non-healing wound, ulcer, or bone fracture.
* If a subject received major surgery, must have recovered adequately from the toxicity and/or complications from the intervention prior to enrollment.
* Clinically significant cardiovascular disease (eg, uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication within 1 year prior to Day -1 (Visit 1); Grade II or greater peripheral vascular disease at study entry
* Any other significant medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study
* History of sensitivity to any component of SD-101
* A diagnosis of cancer within the last 3 years prior to enrollment or any known additional malignancy that is progressing or requires active treatment. Exceptions are B-cell lymphoma, basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, and in situ cervical cancer.
* Is taking systemic corticosteroids (more than 3 consecutive days) or other immunomodulators or immune suppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Leung, MD, Study Director — Dynavax Technologies Corporation
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mooney KL, Czerwinski DK, Shree T, Frank MJ, Haebe S, Martin BA, Testa S, Levy R, Long SR. Serial FNA allows direct sampling of malignant and infiltrating immune cells in patients with B-cell lymphoma receiving immunotherapy. Cancer Cytopathol. 2022 Mar;130(3):231-237. doi: 10.1002/cncy.22531. Epub 2021 Nov 15. PMID 34780125

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg/mL: PART 1: COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29 PART 2: COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29
- 2 mg/mL: PART 1
  COHORT 2: 2 mg/mL at Days 1, 8, 15, 22, and 29
- 4 mg/mL: PART 1
  COHORT 3: 4 mg/mL at Days 1, 8, 15, 22, and 29
- 8 mg/mL: PART 1: COHORT 4: 8 mg/mL at Days 1, 8, 15, 22, and 29 PART 2: COHORT 2: 8 mg/mL at Days 1, 8, 15, 22, and 29
Period: PART 1: Dose Escalation
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Started | 3 | 3 | 3 | 4
Completed | 2 | 0 | 0 | 0
Not Completed | 1 | 3 | 3 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 1 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 3
Not completed — Other | 1 | 1 | 0 | 0
Period: PART 2: Dose Expansion
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Started (Sponsor terminated the trial early during Part 2 and participants should be counted once per row.) | 7 (Participants were enrolled separately from Part 1; sponsor terminated the trial early during Part 2.) | 0 (No new participants were enrolled and sponsor terminated the trial early during Part 2.) | 0 (No new participants were enrolled and sponsor terminated the trial early during Part 2.) | 9 (Participants were enrolled separately from Part 1; sponsor terminated the trial early during Part 2.)
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 9
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 6 | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- 1 mg/mL: PART 1
  COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29
- 8 mg/mL: PART 1
  COHORT 4: 8 mg/mL at Days 1, 8, 15, 22, and 29
- Total: Total of all reporting groups
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL | Total
Number analyzed (Participants) | 10 | 3 | 3 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 2 | 7 | 18
  >=65 years | 3 | 1 | 1 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (13.53) | 56 (9.54) | 61 (16.52) | 62.7 (12.32) | 59.8 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 6 | 13
  Male | 6 | 1 | 2 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 3 | 3 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 3 | 3 | 12 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 3 | 3 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) and Maximum Tolerated Dose (MTD).
Time Frame: Up to Day 36
Population: Safety population
Measure: Number; unit: participants
Groups:
- 1 mg/mL: PART 1: COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29;
  PART 2: COHORT 1: 1 mg/mL at Days 1, 8, 15, 22, and 29
- 8 mg/mL: PART 1: COHORT 4: 8 mg/mL at Days 1, 8, 15, 22, and 29;
  PART 2: COHORT 2: 8 mg/mL at Days 1, 8, 15, 22, and 29
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Number analyzed (Participants) | 10 | 3 | 3 | 13
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: 1 mg/mL vs 2 mg/mL vs 4 mg/mL vs 8 mg/mL; MTD was not observed because no DLTs occurred at the maximum dose tested. Because this is a safety endpoint, a statistical analysis was not conducted; Test type: Other — MTD was not observed because no DLTs occurred at the maximum dose tested. Because this is a safety endpoint, a statistical analysis was not conducted; MTD was not observed because no DLTs occurred at the maximum dose tested. Because this is a safety endpoint, a statistical analysis was not conducted

2. Primary Outcome: Number of Participants Experiencing Injection-site Reactions (ISRs)
Description: Injection site reaction 1 = Redness, Injection site reaction 2 = Swelling, Injection site reaction 3 = Pain
Time Frame: Up to Day 36
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Number analyzed (Participants) | 10 | 3 | 3 | 13
Participants
  Injection site reaction 1 | 4 | 0 | 1 | 5
  Injection site reaction 2 | 4 | 1 | 2 | 2
  Injection site reaction 3 | 7 | 3 | 1 | 6

3. Primary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Time Frame: Up to 38 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Number analyzed (Participants) | 10 | 3 | 3 | 13
participants
  Renal and urinary disorders | 0 | 0 | 0 | 1
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 1 | 0
  Total # of participants with SAEs | 0 | 0 | 1 | 1

4. Primary Outcome: Pharmacodynamic Profile - Expression of IFN-responsive Genes (GBP-1, ISG-54, MCP-1, and MxB)
Description: Fold change of IFN-responsive gene expression relative to Day 8
Time Frame: Change from Day 8 to Day 9
Measure: Geometric Mean (Standard Deviation); unit: Fold Change
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Number analyzed (Participants) | 10 | 3 | 3 | 13
Fold Change | 7.42 (4.78) | 8.06 (2.05) | 9.89 (.59) | 7.78 (7.54)

5. Secondary Outcome: Number of Participants With Preliminary Response - Local (Injected Lesions)
Description: Subjects with maximum decrease of 50% or greater in sum of products of diameters of lesions.
Time Frame: Up to 38 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Number analyzed (Participants) | 9 | 3 | 3 | 13
Participants | 6 | 3 | 1 | 8

6. Secondary Outcome: Number of Participants With Preliminary Response - Systemic (Non-injected Lesions)
Description: Subjects with maximum decrease of 50% or greater in sum of products of diameters of lesions.
Time Frame: Up to 38 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
Number analyzed (Participants) | 9 | 3 | 3 | 13
Participants | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 38 weeks
Arm/Group | 1 mg/mL | 2 mg/mL | 4 mg/mL | 8 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3 | 0/3 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/3 | 1/3 | 1/13
Other Adverse Events (participants affected / at risk) | 10/10 | 3/3 | 3/3 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/mL (N=10) | 2 mg/mL (N=3) | 4 mg/mL (N=3) | 8 mg/mL (N=13)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/mL (N=10) | 2 mg/mL (N=3) | 4 mg/mL (N=3) | 8 mg/mL (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 8
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 5
Asthenia (General disorders) | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 8 | 2 | 3 | 13
Exercise tolerance decreased (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 3 | 3 | 12
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 2
Injection Site Erythema (General disorders) | 4 | 0 | 1 | 3
Injection Site Swelling (General disorders) | 3 | 1 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 2
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 0 | 1
Local swelling (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 9 | 2 | 3 | 13
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 1 | 2 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 0 | 1 | 0 | 0
Dna antibody positive (Investigations) | 0 | 0 | 0 | 1
Eosinophil count decreased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 3 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 8 | 3 | 3 | 11
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cutis laxa (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 2
Hot flush (Vascular disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The sponsor terminated the trial early because there was sufficient data to make a decision about SD-101 in the lymphoma development program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02266147/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT02266147/SAP_001.pdf